CLINICAL TRIAL: NCT00187499
Title: Effect of an Inhaled Corticosteroid on Airway Gene Expression in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Sandler Family Supporting Foundation (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H6788-20160-04; P50HL056385 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2005-09

CONDITIONS: Asthma
Keywords: Asthma; Corticosteroid; Gene expression
MeSH Terms: conditions — Asthma | interventions — BID protein, human

INTERVENTIONS:
Drug: Inhaled fluticasone 500 ug BID for 8 weeks

SUMMARY:
The purpose of this study is to determine whether an inhaled corticosteroid (fluticasone) alters the expression of any gene expressed in the lining of the airways of asthmatics. The study uses high density gene chips which allow the study investigators to measures all gene in the human genome. We hypothesize that this approach will identify novel genes that are affected by steroids in asthmatics.

DETAILED DESCRIPTION:
This is a 10 week, randomized, double blind, prospective study comparing the effects of inhaled fluticasone or inhaled placebo on measures of airway function, airway remodeling and airway gene expression in asthmatic subjects. Enrollment has been completed as have all study visits. We are now in the data analysis phase. The study design was as follows: Following a one-week run-in/characterization period, subjects were randomized to receive 2 puffs BID of fluticasone (250µg/puff) or matching placebo for 8 weeks. Beginning with the run-in period, subjects recordes in a daily diary their peak flow measurements twice daily, (symptoms of cough, sputum production, wheeze, dyspnea, and chest tightness. They visited the laboratory for an interval diary review and spirometry and for medication dispensing. Bronchoscopy was performed at baseline (week 1 of the run-in), and 1 week after starting the study drug Weekly telephone contact will be made during the treatment period to monitor subject well being and to ensure compliance with study medication. There was a one-week run-out to allow monitoring of subjects after discontinuation of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a history of asthma between the ages of 18 and 70 years.
* PC20FEV1 Methacholine ≤ 8.0 mg/mL.
* At least one of the following symptoms, beta agonist use, or FEV1 criteria:
* Asthma symptoms on at least two days per week or Beta agonist use on at least two days per week or FEV1 < 85% predicted
* Subjects must be non-smokers (patients who have never smoked or patients who have not smoked for 1 year and have a total pack-year smoking history < 15 packs).

Exclusion Criteria:

* History of oral or inhaled steroid use in the past 4 weeks.
* FEV1 < 60% predicted.
* Lung disease other than asthma.
* Patients with a history of a respiratory tract infection in the 4 weeks preceding the study.
* Patients who have experienced a significant exacerbation in their asthma in the 6 weeks prior to the study.
* Patients receiving hyposensitization therapy with the exception of those who are on a stable dose for the last three months.
* Patients with cardiovascular disease (active) peptic ulcer disease or diabetes mellitus.
* Females who are lactating or who are pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2005-02

PRIMARY OUTCOMES:
Methacholine responsiveness

SECONDARY OUTCOMES:
gene expression in brushed epithelial cells
lung function

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Airway Clinical Research Center, Room 1303 Moffitt, UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- See also: website for the asthma clinical research group at UCSF — http://allergy.ucsf.edu/